CLINICAL TRIAL: NCT01358799
Title: Clinical Evaluation of the APTIMA® Assay for Chlamydia Trachomatis Using the PANTHER™ System
Status: Withdrawn | Type: Observational
Why Stopped: Assay not evaluated for purpose of clearance
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: ACTPS-US10-001
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Chlamydia Trachomatis
Keywords: Chlamydia trachomatis; APTIMA Assay for Chlamydia trachomatis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 4 specimens will be collected from each female subject in the following order: 1 first-catch urine specimen, 1 vaginal swab specimen (patient or clinician-collected), 1 cervical specimen (using a broomlike collection device or a brush/spatula combination), and 1 endocervical swab specimen. An additional cervical specimen may be collected from female subjects for other clinical trial purposes or research studies. Up to 2 specimens will be collected from each male subject in the following order: 1 urethral swab specimen and 1 first-catch urine specimen.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: APTIMA Assay for Chlamydia trachomatis — APTIMA Assay for Chlamydia trachomatis
  Other Names: Chlamydia trachomatis

SUMMARY:
The objective of this multi-center clinical study is to demonstrate that the APTIMA(R) Assay for Chlamydia trachomatis (CT; "ACT Assay"), which is cleared for use on the TIGRIS DTS (Direct Transfer) System ("TIGRIS System"), can be tested on the PANTHER System. The intended use of the ACT Assay will be unchanged except for the inclusion of its use with the PANTHER System. ACT Assay performance on the PANTHER System is comparable to performance on the TIGRIS System.

DETAILED DESCRIPTION:
This protocol was withdrawn from clinical trials.gov because samples collected under this protocol were not tested per protocol using the Gen-Probe APTIMA(R) CT (Chlamydia trachomatis) Assay. Instead, testing was conducted and results were generated with the Gen-Probe APTIMA(R) Combo 2 Assay (for Chlamydia trachomatis and Neisseria gonorrhoeae). See Protocol Identification AC2PS-US11-001 (NCT01733069) for results. This action was recommended by the RRS team per their email to me on 8 February 2013.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 14 years of age at the time of informed consent and is sexually active

  * The subject reports symptoms consistent with a suspected STD such as abnormal discharge, genital itching, pain/discomfort during sexual intercourse or urination, and/or lower abdominal discomfort.
  * If the subject is asymptomatic, the subject is known to be partners with, or a contact of, a person with a confirmed or suspected STD(s), is undergoing screening evaluation for a possible STD(s), and/or is scheduled for a routine exam that may include a pelvic exam
  * The subject and/or legally authorized representative is willing to undergo the informed consent process prior to study participation (a minor will need the documented consent of his/her parent or legal guardian, unless the site has an IRBapproved waiver for parental consent for minors)

Exclusion Criteria:

* A potential subject will be ineligible for clinical trial enrollment if the subject, clinician, or medical record reports any of the following:

  * The subject took antibiotic medications within the last 21 days
  * The subject is underage (as defined by the IRB or state law), without the documented consent of her/his parent or legal guardian (exception: sites that have an IRBapproved waiver for parental consent for minors)
  * The subject is determined by the investigator to be medically unsuitable for participation in this study (eg, medical history of concurrent illness that could result in an unacceptable risk to the subject) Concurrent participation in other clinical study(ies) may be acceptable, with approval by the investigator and sponsor.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male and Females at least 14 years of age at the time of informed consent and sexually active.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Percent Agreement Using the TIGRIS Instrument as a Reference | approximately one year
  Positive and Negative Percent Agreement Using the TIGRIS Instrument as a Reference

SECONDARY OUTCOMES:
Positivity Rate | approximately one year
  Positivity Rate

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reid, PhD, Study Director — Gen-Probe, Incorporated
Locations (7):
- United States (7):
  - Wishard Health Services Department of Pathology Wishard Health Services, Indianapolis, Indiana
  - Louisianna State University Health Center, New Orleans, Louisiana
  - New England Center for Clinical Research, Fall River, Massachusetts
  - University of North Carolina Chapel Hill STD Clinic, Chapel Hill, North Carolina
  - Planned Parenthood Northeast Ohio, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center Division of Pediatric & Adolescent Gynecology, Cincinnati, Ohio
  - Planned Parenthood Houston and Southeast Texas, Houston, Texas